CLINICAL TRIAL: NCT03333148
Title: Preoperative Oral ImmunoNuTrition to Improve Surgical Outcomes for Inflammatory Bowel Disease Patients (PINT): A Randomized Controlled Trial
Brief Title: Preoperative Oral ImmunoNuTrition to Improve Surgical Outcomes for IBD Patients (PINT)
Acronym: PINT
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: never enrolled
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gregory D. Kennedy, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB -170222002
Record Dates: First submitted 2017-10-20; First posted 2017-11-06 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Colorectal Surgery; Immunonutrition; Complications; Microbiome; Preoperative nutrition
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - Nestle IMPACT Immunonutrition (Experimental): Treatment Arm A (n=146) - Nestlé IMPACT Advanced Recovery:Along with standard of care nutritional therapy patients will be asked to consume 3 cartons/day for 14 days of Nestle IMPACT Advanced Recovery Immunonutrition.
  Interventions: Drug: Nestle IMPACT Immunonutrition
- Arm B- Standard of Care (Other): No intervention standard of care nutrition (n=146).
  Interventions: Other: Arm B- Standard of Care

INTERVENTIONS:
Drug: Nestle IMPACT Immunonutrition — Along with standard of care nutritional therapy patients (n=146) will be asked to consume 3 cartons/day for 14 days of Nestle IMPACT Advanced Recovery Immunonutrition.
  Other Names: Nestle IMPACT Advanced Recovery Immunonutrition
  Arms: Arm A - Nestle IMPACT Immunonutrition
Other: Arm B- Standard of Care — No intervention standard of care nutrition (n=146).
  Other Names: Standard of Care
  Arms: Arm B- Standard of Care

SUMMARY:
The central focus of this trial is to understand the effectiveness of Preoperative Immunonutrition (PINT) in improving surgical outcomes for patients with inflammatory bowel disease (IBD). We hypothesize that PINT will reduce post-operative complications in IBD patients undergoing elective surgery with added improvements in length-of-stay (LOS), quality of life (QOL) and patient satisfaction. As a secondary focus, the investigator will aim to better understand the potential mechanism-of-action by which PINT may have its effects through analyses of biomarkers including inflammatory markers, nutritional proteins and the fecal microbiome.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD), which includes Crohn's and Ulcerative Colitis, is a chronic and costly disease of unknown etiology that now affects over 3.1 million people in the United States. Patients with IBD suffer from lifelong malnutrition, pain and bleeding with added risks of cancers, obstructions and fistulas. There is no known cure and the incidence continues to grow. While treatments are usually medical IBD patients will undergo at least one major surgery during their lifetime. Patients also have particularly poor surgical outcomes with high rates of post-operative complications. In an attempt to improve the risk profile of patients and decrease complications, preoperative total parenteral nutrition (TPN) has been used to optimize IBD patients for surgery. While this approach has been successful the cost and morbidities of TPN prohibit its generalized application. Practical strategies that improve surgical outcomes for IBD patients are urgently needed. Improving nutritional deficiencies before an operation may be a practical way to improve post-operative outcomes. The oral administration of preoperative immunonutrition, is an alternative method to improve nutritional states and may have utility in IBD patients who have particularly severe nutritional deficiencies because of disease-specific issues in malabsorption, maldigestion and loss of appetite.

ELIGIBILITY:
Inclusion Criteria:

* ≥19 years of age
* All races and all genders
* Confirmed diagnosis and history of IBD
* ESPEN Nutritional Risk Scores >=3 and the ESPEN Disease Severity sub-score < 3
* Scheduled for elective surgery via any transabdominal operative approach (i.e. laparoscopic, hand-assisted, robotic, open) with a planned postoperative inpatient stay of at least one night

Exclusion Criteria:

* Failure to meet eligibility criteria
* Patients requiring emergency surgical intervention
* Patients with an American Society of Anesthesiologist physical status of IV or V
* Patients requiring hemodialysis
* Patients with history of myocardial infarction within 6 months
* Patients with a history of asthma
* Patients with cirrhosis or a history of liver disease
* Patients with a present history of dysphagia, pyloric stenosis and esophageal strictures
* Patients unable to consume liquids orally
* Patients allergic or with hypersensitivity reactions to any of the components of the Nestlé IMPACT-Advanced Recovery immunonutritional supplement
* Patients with a history of galactosemia, the inability to metabolize the sugar galactose appropriately
* Patients with bowel obstructions
* Patients with history of HIV or of solid-organ transplant
* Patients who are pregnant or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
The occurrence of any postoperative complications after surgery | Baseline (day of surgery) to 2 weeks (after surgery)
  Routine postoperative follow-up for all patients will occur at 2 weeks post discharge. Any serious adverse events or adverse events will be ascertained at the 2 week follow up visit. Complication rates will be divided into major and minor postoperative complications and will be defined as any deviation from the normal postoperative recovery process. Complications will be assessed using the Clavien-Dindo classification in minor and major.
The occurrence of any postoperative complications after surgery | Baseline (day of surgery) to 30 days (after surgery)
  At the 30 day post-discharge postoperative follow up visit, serious adverse events will be ascertained that may have occurred after the 2 week follow up visit. Patients who are unable to return on the 30-day mark will be called to screen for any post-discharge complications. Complication rates will be divided into major and minor postoperative complications and will be defined as any deviation from the normal postoperative recovery process. Complications will be assessed using the Clavien-Dindo classification in minor and major.
The occurrence of any postoperative complications after surgery | Baseline (day of surgery) to 60 days (after surgery)
  Final call to ascertain complications will be at 60 days. Complication rates will be divided into major and minor postoperative complications and will be defined as any deviation from the normal postoperative recovery process. Complications will be assessed using the Clavien-Dindo classification in minor and major.

SECONDARY OUTCOMES:
Detection of the differences in the markers of inflammation interleukin-1-β (IL-1β) | Baseline (preoperative visit)
  Enzyme-linked immunosorbent assays (ELISA) will be performed to assess whole blood, plasma and serum samples for circulating inflammatory cytokine interleukin-1-β (IL-1β.
Detection of the differences in the markers of inflammation interleukin-1-β (IL-1β) | Baseline (preoperative visit) to day of surgery
  Enzyme-linked immunosorbent assays (ELISA) will be performed to assess whole blood, plasma and serum samples for circulating inflammatory cytokine interleukin-1-β (IL-1β.
Detection of the differences in the markers of inflammation interleukin-1-β (IL-1β) | Baseline (preoperative visit) to postoperative day 3
  Enzyme-linked immunosorbent assays (ELISA) will be performed to assess whole blood, plasma and serum samples for circulating inflammatory cytokine interleukin-1-β (IL-1β.
Detection of the differences in the markers of inflammation Interleukin 6 (IL-6) | Baseline (preoperative visit)
  Enzyme-linked immunosorbent assays (ELISA) will be performed to assess whole blood, plasma and serum samples for circulating inflammatory cytokine interleukin-6 (IL-6).
Detection of the differences in the markers of inflammation Interleukin 6 (IL-6) | Baseline (preoperative visit) to day of surgery
  Enzyme-linked immunosorbent assays (ELISA) will be performed to assess whole blood, plasma and serum samples for circulating inflammatory cytokine interleukin-6 (IL-6).
Detection of the differences in the markers of inflammation Interleukin 6 (IL-6) | Baseline (preoperative visit) to postoperative day 3
  Enzyme-linked immunosorbent assays (ELISA) will be performed to assess whole blood, plasma and serum samples for circulating inflammatory cytokine interleukin-6 (IL-6).
Detection of the differences in the markers of inflammation tumor necrosis factor (TNF-α) | Baseline (preoperative visit)
  Enzyme-linked immunosorbent assays (ELISA) will be performed to assess whole blood, plasma and serum samples for circulating tumor necrosis factor (TNF-α).
Detection of the differences in the markers of inflammation tumor necrosis factor (TNF-α) | Baseline to day of surgery
  Enzyme-linked immunosorbent assays (ELISA) will be performed to assess whole blood, plasma and serum samples for circulating tumor necrosis factor (TNF-α).
Detection of the differences in the markers of inflammation tumor necrosis factor (TNF-α) | Baseline (preoperative visit) to postoperative day 3
  Enzyme-linked immunosorbent assays (ELISA) will be performed to assess whole blood, plasma and serum samples for circulating tumor necrosis factor (TNF-α).
Detection of the differences in the markers of inflammation CRP | Baseline (preoperative visit)
  Immunoassays will be performed with high sensitivity nephelometry to measure CRP levels.
Detection of the differences in the markers of inflammation CRP | Baseline (preoperative visit) to day of surgery
  Immunoassays will be performed with high sensitivity nephelometry to measure CRP levels.
Detection of the differences in the markers of inflammation CRP | Baseline (preoperative visit) to postoperative day 3
  Immunoassays will be performed with high sensitivity nephelometry to measure CRP levels.
Detection of the differences in the markers of inflammation nutritional status albumin | Baseline (preoperative visit)
  Comprehensive metabolic panels will be ordered to assess levels of serum albumin
Detection of the differences in the markers of inflammation nutritional status albumin | Baseline (preoperative visit) to day of surgery
  Comprehensive metabolic panels will be ordered to assess levels of serum albumin
Detection of the differences in the markers of inflammation nutritional status albumin | Baseline (preoperative visit) to postoperative day 3
  Comprehensive metabolic panels will be ordered to assess levels of serum albumin
Detection of the differences in the markers of inflammation pre-albumin | Baseline (preoperative visit)
  Comprehensive metabolic panels will be ordered to assess levels of serum pre-albumin
Detection of the differences in the markers of inflammation pre-albumin | Baseline (preoperative visit) to day of surgery
  Comprehensive metabolic panels will be ordered to assess levels of serum pre-albumin
Detection of the differences in the markers of inflammation pre-albumin | Baseline (preoperative visit) to postoperative day 3
  Comprehensive metabolic panels will be ordered to assess levels of serum pre-albumin

OTHER OUTCOMES:
Length of hospital stay (LOS) | Baseline (Day of surgery) to day of discharge (approximately 2 to 30 days post surgery)
  Length of stay will be captured through patient hospitalization files
Patient Quality of Life (QOL) | Baseline (preoperative visit)
  At the time of the pre-operative visit, following enrollment in the study, participants will complete the Health Related Quality of Life Survey SF-12 questionnaire (HRQoL SF-12). The results of the Health Related Quality of Life Survey SF-12 questionnaire (HRQoL SF-12) will be analyzed and Physical and Mental Health Composite Scores (PCS & MCS) will be computed using the scores of the twelve questions ranging from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Patient Quality of Life (QOL) | Baseline (preoperative) to 30 days
  Patients at their two week follow up postoperative visit will be given another copy of the HRQoL SF-12 and prepaid return envelopes to be completed and mailed back two weeks after follow up Patients will receive a reminder call to complete the surveys and return in the mail. The results of the Health Related Quality of Life Survey SF-12 questionnaire (HRQoL SF-12) will be analyzed and Physical and Mental Health Composite Scores (PCS & MCS) will be computed using the scores of the twelve questions ranging from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Patient Satisfaction (S-CAHPS) | Baseline (Preoperative)
  Will be captured preoperatively with the S-CAHPS. Participants will be asked to complete the Surgical-Consumer Assessment of Healthcare Providers and Systems (S-CAHPS) Survey. The S-CAHPS Surgical Care Survey was developed in 2009 through collaboration of the CAHPS consortium, American College of Surgeons (ACS), the Surgical Quality Alliance (SQA), the American Urological Association (AUA), 11 other surgical subspecialty groups and endorsed by the National Quality Forum (NQF) in 2012. The S-CAHPS is a 47 question survey that addresses patients' preoperative and postoperative experience with surgical care. The CAHPS Surgical Care Survey generates a global rating item, which uses a scale of 0 to 10 to measure respondents' assessments of their surgeon and composite measures (also known as reporting composites), which combine results for closely-related items that have been grouped together.
Patient Satisfaction (S-CAHPS) | Postoperative (After Surgery)
  Will be captured postoperatively with the S-CAHPS. Participants will be asked to complete the Surgical-Consumer Assessment of Healthcare Providers and Systems (S-CAHPS) Survey. The S-CAHPS Surgical Care Survey was developed in 2009 through collaboration of the CAHPS consortium, American College of Surgeons (ACS), the Surgical Quality Alliance (SQA), the American Urological Association (AUA), 11 other surgical subspecialty groups and endorsed by the National Quality Forum (NQF) in 2012. The S-CAHPS is a 47 question survey that addresses patients' preoperative and postoperative experience with surgical care. The CAHPS Surgical Care Survey generates a global rating item, which uses a scale of 0 to 10 to measure respondents' assessments of their surgeon and composite measures (also known as reporting composites), which combine results for closely-related items that have been grouped together.
Detection of differences in fecal microbiome | Baseline (Preoperative)
  For fecal microbiome analyses, stool will be processed for 16S rRNA sequencing. DNA will be extracted from stool samples using the Fecal DNA Isolation Kit (Zymo Research, Irvine, CA) and processed with PCR amplification on the MiSeq. QIIME and UniFrac will be used to generate a comparative profile of microbial composition. QIIME will be used to assess taxa, alpha and beta diversity. Composition of the microbiome will be compared using UniFrac, Mothur and Genboree to assess for differences between microbiome populations by principal components analysis.
Detection of differences in fecal microbiome | Day of Surgery
  For fecal microbiome analyses, stool will be processed for 16S rRNA sequencing. DNA will be extracted from stool samples using the Fecal DNA Isolation Kit (Zymo Research, Irvine, CA) and processed with PCR amplification on the MiSeq. QIIME and UniFrac will be used to generate a comparative profile of microbial composition. QIIME will be used to assess taxa, alpha and beta diversity. Composition of the microbiome will be compared using UniFrac, Mothur and Genboree to assess for differences between microbiome populations by principal components analysis.
Detection of differences in fecal microbiome | 2 weeks after surgery (postoperative visit)
  For fecal microbiome analyses, stool will be processed for 16S rRNA sequencing. DNA will be extracted from stool samples using the Fecal DNA Isolation Kit (Zymo Research, Irvine, CA) and processed with PCR amplification on the MiSeq. QIIME and UniFrac will be used to generate a comparative profile of microbial composition. QIIME will be used to assess taxa, alpha and beta diversity. Composition of the microbiome will be compared using UniFrac, Mothur and Genboree to assess for differences between microbiome populations by principal components analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Kennedy, MD,PhD, Principal Investigator — University of Alabama at Birmingham